CLINICAL TRIAL: NCT04992507
Title: The Impact of Total Intravenous Anesthesia Following Cancer Surgery (TIVACS) Study
Brief Title: Impact of Total Intravenous Anesthesia Following Cancer Surgery, TIVACS Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator departed sponsoring organization
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20306; NCI-2021-05849 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Anesthesia; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (surgical resection with TIVA) (Experimental): Patients undergo surgical resection with TIVA.
  Interventions: Procedure: Anesthesia Procedure; Procedure: Resection
- Arm II (surgical resection with inhaled volatile anesthetics) (Active Comparator): Patients undergo surgical resection with inhaled volatile anesthetics.
  Interventions: Drug: General Anesthesia Procedure; Procedure: Resection

INTERVENTIONS:
Procedure: Anesthesia Procedure — Given TIVA
  Other Names: Anesthesia
  Arms: Arm I (surgical resection with TIVA)
Drug: General Anesthesia Procedure — Given inhaled volatile anesthetics
  Other Names: General Anesthesia
  Arms: Arm II (surgical resection with inhaled volatile anesthetics)
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection

SUMMARY:
This phase II trials studies the impact of total intravenous anesthesia (TIVA) following cancer surgery. Surgery and the anesthesia delivered causes physiologic stress and trauma resulting in immune suppression. TIVA is an alternative method of general anesthesia that has several benefits over volatile inhalation agents such as reducing nausea, vomiting, and opioid consumption, and promotes earlier return of bowel function following surgery. In addition, TIVA is less immunosuppressive than inhalational agents and has been shown to decrease cancer cell proliferation, migration, and metastasis formation. Giving TIVA during cancer-directed abdominal surgery may decrease the immunosuppressive state in the peri-surgical period.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the impact of anesthetic agent on inflammation and immunosuppression among patients undergoing abdominal cancer surgery.

SECONDARY OBJECTIVE:

I. To determine the impact of anesthetic choice on short-term anesthetic and surgical outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo surgical resection with TIVA.

ARM II: Patients undergo surgical resection with inhaled volatile anesthetics.

After completion of study treatment, patients are followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults: ≥18 years old on the day of consent
* Non-metastatic pancreatic adenocarcinoma
* Able to provide consent
* ECOG performance status of 0 or 1
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test for the patient at the time of surgery.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Previous identified allergy or hypersensitivity to any component of the study treatment
* Allergies to eggs, egg products, soybeans, or soy products
* Personal or first degree relative with a history of malignant hyperthermia
* Has a known additional malignancy that is expected to require active treatment within two years, or is likely to be life-limiting in the opinion of the treating investigator. Superficial bladder cancer, non-melanoma skin cancers, or low-grade prostate cancer not requiring therapy would not exclude participation in this trial.
* Uncontrolled intercurrent illness including, but not limited to: Symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating females
* Major surgery within 2 months before enrollment. Complete healing from major surgery must have occurred 1 month before enrollment. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before enrollment. Subjects with clinically relevant complications from prior surgery are not eligible.

  * Patients who undergo reoperation during their initial hospitalization will be censored at the time of reoperation.
* Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aslam Ejaz, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Surgical Resection With TIVA) | Arm II (Surgical Resection With Inhaled Volatile Anesthetics)
Started | 5 | 3
Treatment | 1 | 0
Completed | 0 | 0
Not Completed | 5 | 3
Not completed — Study terminated early due to principal investigator departing sponsoring organization | 5 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Surgical Resection With TIVA) | Arm II (Surgical Resection With Inhaled Volatile Anesthetics) | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Impact of Anesthetic Agent on Inflammation and Immunosuppression
Description: All data analysis will use Student's t-test, Chi2 test and multivariable regression analysis using linear mixed model. The incidence of these outcomes will also be associated with NET levels.
Time Frame: Up to 2 years
Population: Due to the early termination of the study, only one participant underwent surgery and received treatment and that participant did not stay on study long enough to have data collected for the primary or secondary outcome measure. Therefore, there is no collected data to report for this outcome measure.
Arm/Group | Arm I (Surgical Resection With TIVA) | Arm II (Surgical Resection With Inhaled Volatile Anesthetics)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Impact of Anesthetic Choice on Short-term Anesthetic and Surgical Outcomes
Description: as for outcome 1
Time Frame: Up to 2 years
Population: as for outcome 1
Arm/Group | Arm I (Surgical Resection With TIVA) | Arm II (Surgical Resection With Inhaled Volatile Anesthetics)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline until the study was terminated, an average of 1.5 months for each participant
Arm/Group | Arm I (Surgical Resection With TIVA) | Arm II (Surgical Resection With Inhaled Volatile Anesthetics)
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 3/5 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Surgical Resection With TIVA) (N=5) | Arm II (Surgical Resection With Inhaled Volatile Anesthetics) (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT04992507/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT04992507/ICF_001.pdf